CLINICAL TRIAL: NCT00000371
Title: A Six Month, Placebo-Controlled Trial of D-Cycloserine Co-Administered With Conventional Antipsychotics in Schizophrenia Patients
Brief Title: Trial of D-Cycloserine in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH054245-01A2 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Adult; Cognition; Cycloserine; Dopamine; Female; Glutamic Acid; Human; Male; Receptors, N-Methyl-D-Aspartate; Schizophrenia; Serotonin; Quality of Life; Cycloserine -- *therapeutic use; Dopamine -- blood; Dopamine -- cerebrospinal fluid; Glutamic Acid -- blood; Glutamic Acid -- cerebrospinal fluid; Serotonin -- blood; Serotonin -- cerebrospinal fluid
MeSH Terms: conditions — Schizophrenia | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- D-Cycloserine (Experimental): Subjects were given 50 mg/day of D-Cycloserine for 24 weeks
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator): Participants were given 50 mg/day of Placebo for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg/daily by mouth
  Other Names: Cycloserine
  Arms: D-Cycloserine
Drug: Placebo — 50 mg/day of placebo by mouth
  Arms: Placebo

SUMMARY:
To characterize further the effects of D-cycloserine augmentation of antipsychotic treatment on negative symptoms, performance on neurocognitive tasks, and on markers for glutamatergic, dopaminergic and serotonergic function in serum and cerebrospinal fluid. To determine if negative symptoms and cognitive function improve over time, if these improvements meaningfully impact quality of life factors, if they correlate with markers of neuronal function, and if subpopulations can be identified according to response.

Dysfunction of glutamatergic neuronal systems has recently been implicated in the pathophysiology of schizophrenia based on the finding that non-competitive inhibitors of the NMDA receptor can reproduce in normals the positive symptoms, negative symptoms, and cognitive deficits of schizophrenia. Furthermore, glutamatergic dysfunction may alter forebrain dopaminergic neuronal activity, a system central to the antipsychotic action of typical neuroleptics. It is believed that enhancing NMDA receptor function by systemic treatment with D-cycloserine, a partial agonist at the glycine modulatory site of the NMDA receptor, will reduce symptoms in schizophrenia.

Sixty schizophrenic outpatients with prominent, primary negative symptoms are treated with antipsychotic medication and are randomly assigned to D-cycloserine or placebo for a 6-month, fixed-dose trial. The primary outcome measure is the total score on the Scale for Assessment of Negative Symptoms (SANS). A neuropsychological battery, which emphasizes tests sensitive to prefrontal cortical function, is administered. Blood is obtained at several time points and CSF is obtained at Week 8 for assay of concentrations of D-cycloserine, glutamate, HVA, and 5HIAA.

DETAILED DESCRIPTION:
To characterize further the effects of D-cycloserine augmentation of antipsychotic treatment on negative symptoms, performance on neurocognitive tasks, and on markers for glutamatergic, dopaminergic, and serotonergic function in serum and cerebrospinal fluid. To determine if negative symptoms and cognitive function improve over time, if these improvements meaningfully impact quality of life factors, if they correlate with markers of neuronal function, and if subpopulations can be identified according to response.

Dysfunction of glutamatergic neuronal systems has recently been implicated in the pathophysiology of schizophrenia based on the finding that non-competitive inhibitors of the NMDA receptor can reproduce in normals the positive symptoms, negative symptoms and cognitive deficits of schizophrenia. Furthermore, glutamatergic dysfunction may alter forebrain dopaminergic neuronal activity, a system central to the antipsychotic action of typical neuroleptics. It is believed that enhancing NMDA receptor function by systemic treatment with D-cycloserine, a partial agonist at the glycine modulatory site of the NMDA receptor, will reduce symptoms in schizophrenia.

Sixty schizophrenic outpatients with prominent, primary negative symptoms are treated with antipsychotic medication and are randomly assigned to D-cycloserine or placebo for a 6-month, fixed-dose trial. The primary outcome measure is the total score on the Scale for Assessment of Negative Symptoms (SANS). A neuropsychological battery, which emphasizes tests sensitive to prefrontal cortical function, is administered. Blood is obtained at several time points and CSF is obtained at Week 8 for assay of concentrations of D-cycloserine, glutamate, HVA, and 5HIAA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia as per DSM IV criteria
* Have been treated for at least 6 months with any conventional neuroleptic
* Have prominent negative symptoms as defined by a total score of 40 or greater on the scale for the assessment of negative symptoms (SANS)

Exclusion Criteria:

* Active alcohol or drug abuse
* Unstable Medical Illness, seizure disorder, or other serious neurological disorder
* Pregnant or Nursing
* Unable to complete a cognitive battery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1996-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator

REFERENCES:
- [Result] Goff DC, Herz L, Posever T, Shih V, Tsai G, Henderson DC, Freudenreich O, Evins AE, Yovel I, Zhang H, Schoenfeld D. A six-month, placebo-controlled trial of D-cycloserine co-administered with conventional antipsychotics in schizophrenia patients. Psychopharmacology (Berl). 2005 Apr;179(1):144-50. doi: 10.1007/s00213-004-2032-2. Epub 2004 Oct 21. PMID 15502972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were adult outpatients recruited from three urban community health centers and two Veteran's Affairs medical centers in the greater Boston area. All eligible participants at these sites were invited to participate by their clinicians.
Pre-assignment Details: Sixty subjects met eligibility criteria and provided informed consent, but just 55 completed baseline assessments and were randomized to d-cycloserine or placebo.
Groups:
- D-Cycloserine: Patients were given 50 mg of D-Cycloserine daily in addition to their treatment as usual with conventional neuroleptics.
- Placebo: Patients were given 50 mg of placebo daily in addition to their treatment as usual with conventional neuroleptics.
Period: Overall Study
Arm/Group | D-Cycloserine | Placebo
Started | 27 | 28
Completed | 14 | 12
Not Completed | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-Cycloserine | Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (7.4) | 47.0 (8.6) | 46.5 (8.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 24 | 20 | 44
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: The slope of SANS total score from baseline to week 8 in the treatment and placebo groups on the scale for the assessment of negative symptoms (SANS) total score. Total SANS scores range from 0-100. The SANS is comprised of 5 subscores: Affective Flattening or Blunting (score range 0-35), Alogia (score range 0-20), Avolition-Apathy (score range 0-15), Anhedonia-Asociality (score range 0-20), and Attention (0-10). For each scale, the higher the score the more prominent the negative symptoms were. The slopes were obtained by plotting the group SANS total score mean for treatment vs. placebo on Baseline, Week 4, and Week 8 and performing a random slopes model.
Time Frame: Baseline, Week 4, Week 8
Measure: Mean (Standard Error); unit: units on a scale/weeks
Arm/Group | D-Cycloserine | Placebo
Number analyzed (Participants) | 28 | 27
units on a scale/weeks | -.46 (.29) | -.41 (.31)

ADVERSE EVENTS:
Description: The only information known for this study regarding occurrence of Adverse Events is that 2 and 6 participants dropped out of the D-Cycloserine and Placebo Arms/Groups, respectively (reported in the publication associated with this clinical trials profile). However, specific adverse event data are lost and cannot be retrieved
Arm/Group | D-Cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A biased sample may have been produced by restricting the analysis to patients with prominent negative symptoms receiving conventional agents (less compliant with study medication). Additionally, Adverse Event data was lost for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No